CLINICAL TRIAL: NCT05440955
Title: Efficacy and Auditory Biomarker Analysis of Fronto-Temporal Transcranial Direct Current Stimulation (tDCS) in Targeting Cognitive Impairment Associated With Recent-onset Schizophrenia: A Randomized Double-blind Sham-controlled Trial
Brief Title: tDCS for Cognitive Impairment Associated With Recent-onset Schizophrenia
Acronym: STICOG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STICOG
Record Dates: First submitted 2022-05-31; First posted 2022-07-01 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenia; Psychotic Disorder
Keywords: schizophrenia; cognitive impairment; tDCS; early auditory processing; clinical trial
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The present study is designed as a superiority, double-blind, parallel-group, sham-controlled randomized clinical trial with an allocation ratio of 1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be maintained at several levels: participants, research staff members including investigators and data analysts. If different from the investigator, care providers will be also blinded to intervention. Blinding for the tDCS condition will be achieved for the research staff members who will administer the tDCS by the use of a randomization code (see details in §16c) and for the participants by ensuring identical appearance and sensation for both active and sham conditions. Outcome assessments, imaging and biological data will be collected and analysed by research staff members blind to group assignment and different from the staff member who will administer the tDCS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Experimental): tDCS (transcranial Direct Current Stimulation subjects) is a noninvasive brain stimulation technique that involves the passage of a small electric current through the scalp and skull to modulate brain activity [10]. The study intervention consists of ten 20-minutes sessions of active or sham tDCS. Sessions will be delivered twice daily and separated by at least 2 hours for 5 consecutive weekdays. The electric current will be generated by an electric stimulator (class IIa medical device).
  Interventions: Device: left fronto-temporal transcranial Direct Current Stimulation (tDCS)
- sham tDCS (Sham Comparator): The sham procedure is developed by the tDCS device manufacturer, which allows using the same tDCS device and the same procedure (i.e., 10 sessions delivered during five consecutive days) for both the active and sham procedures. In the sham condition, the electrodes will be placed in the same positions as in the active group; however, the stimulator will be only active for initial and final ramp up/ramp down periods, in order to mimic the sensation of active stimulation. In addition, brief pulses of 110 μA will be administered every 550 ms in order to control impedance and keep the manipulator blinded to the active or sham condition.
  Interventions: Device: left fronto-temporal transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: left fronto-temporal transcranial Direct Current Stimulation (tDCS) — The study intervention consists of ten 20-minutes sessions of active or sham tDCS. Sessions will be delivered twice daily and separated by at least 2 hours for 5 consecutive weekdays. The electric current will be generated by an electric stimulator (class IIa medical device). During the entire tDCS session, the subject is at "rest", comfortably seated in a chair in a quiet room. A clinician will be present for the entire session duration. The current will be applied via a pair of rubber electrodes (35 cm²) placed on the surface of the scalp. The anode will be placed over the left dorsolateral prefrontal cortex. The cathode will be placed over the left auditory cortex. The stimulation parameters will be set at 2-mA for 20 minutes, with a progressive increase during the first 30-sec and a progressive decrease during the last 30-sec of each session. The impedance of the applied current is monitored by the stimulator during each session.

SUMMARY:
Background: In parallel to the traditional symptomatology, deficits in cognition (memory, attention, reasoning, social functioning) contribute significantly to disability and suffering in individuals with schizophrenia. Cognitive deficits have been closely linked to alterations in early auditory processes (EAP) that occur in auditory cortical areas. Preliminary evidence indicates that cognitive deficits in schizophrenia can be improved with a reliable and safe non-invasive brain stimulation technique called tDCS (transcranial Direct Current Stimulation). However, a significant proportion of patients derive no cognitive benefits after tDCS treatment. Further, the neurobiological mechanisms of cognitive changes after tDCS have been poorly explored in trials and are thus still unclear.

Method: The study is designed as a randomized, double-blind, 2-arm parallel-group, sham controlled, 4-centers trial. Sixty participants with recent-onset schizophrenia and cognitive impairment will be randomly allocated to receive either active (n=30) or sham (n=30) tDCS (20-min, 2-mA, 10 sessions during 5 consecutive weekdays). The anode will be placed over the left dorsolateral prefrontal cortex and the cathode over the left auditory cortex. Cognition, tolerance, symptoms, general outcome and EAP (measured with EEG and multimodal MRI) will be assessed prior to tDCS (baseline), after the 10 sessions, and at 1- and 3-month follow-up. The primary outcome will be the number of responders, defined as participants demonstrating a cognitive improvement ≥Z=0.5 from baseline on the MATRICS Consensus Cognitive Battery total score at 1-month follow-up. Additionally, we will measure how differences in EAP modulate individual cognitive benefits from active tDCS and whether there are changes in EAP measures in responders after active tDCS.

Discussion: Besides proposing a new fronto-temporal tDCS protocol by targeting the auditory cortical areas, we aim to conduct an RCT with follow-up assessments up to 3-months and a large sample size. In addition, this study will allow identifying and assessing the value of a wide range of neurobiological EAP measures for predicting and explaining cognitive deficits improvement after tDCS. The results of this trial will constitute a step toward the use of tDCS as a therapeutic tool for the treatment of cognitive impairment in recent-onset schizophrenia.

ELIGIBILITY:
The inclusion criteria include:

1. subjects of both genders, diagnosed with recent-onset schizophrenia (first 3 years of illness), confirmed through the Structured Clinical Interview for the American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders, 5th edition (SCID-5);
2. aged 18-35 years;
3. intelligence quotient (IQ) > 55;
4. cognitive deficit confirmed by a MCCB (MATRICS Cognitive Consensus Battery) total score T-score < 40;
5. the subjects should be receiving stable doses of antipsychotics for ≥ 4 weeks;
6. the subjects are covered by a public health insurance.

The exclusion criteria include:

1. pregnant (controlled by urine pregnancy test in females of childbearing age) or breastfeeding women;
2. unstable or acute medical conditions;
3. subjects who receive involuntary treatment or guardianship;
4. history of cranioencephalic trauma with loss of consciousness or central nervous system diseases that affect the brain;
5. use of drugs that affect cognitive performance such as anticholinergic agents and benzodiazepines;
6. current diagnosis of substance abuse or history of substance dependence in the last 6 months, except nicotine;
7. MRI (Magnetic Resonance Imaging), PET (Positron Emission Tomography) or tDCS (transcranial Direct Current Stimulation) contraindications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive response | at 1-month follow-up
  Number of responders at 1-month after tDCS, defined as the proportion of patients demonstrating a cognitive improvement greater than or equal to Z=0.5 from baseline on the MATRICS Consensus Cognitive Battery total score (MCCB). The MCCB is a gold-standard standardized test battery to assess cognitive functions in patients with schizophrenia. This criterion has been used and validated in both antipsychotic and cognitive remediation trials in schizophrenia.

SECONDARY OUTCOMES:
Long term cognitive response | at inclusion; at 3-months follow-up
  Number of responders at 3-months after tDCS, defined as the proportion of patients demonstrating a cognitive improvement greater than or equal to Z=0.5 from baseline on the MATRICS Consensus Cognitive Battery total score (MCCB). The MCCB is a gold-standard standardized test battery to assess cognitive functions in patients with schizophrenia. This criterion has been used and validated in both antipsychotic and cognitive remediation trials in schizophrenia.
Cognitive domain response | at inclusion; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to 1-month and 3-months endpoints in each MCCB domains subscores (processing speed, attention/vigilance, working memory, verbal learning, visual learning, problem solving, emotional awareness) and total score.
Clinical response 1 | at inclusion; at 1-week; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to after tDCS, 1-month and 3-months endpoints in the following symptom measure:
  • Schizophrenia symptoms will be assessed using the PANSS (Positive and Negative Syndrome Scale) total score.
Clinical response 2 | at inclusion; at 1-week; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to after tDCS, 1-month and 3-months endpoints in the following symptom measure:
  • Auditory hallucinations, one of the key symptoms of schizophrenia, will be assessed using the AHRS (Auditory Hallucination Rating Scale)
Clinical response 3 | at inclusion; at 1-week; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to after tDCS, 1-month and 3-months endpoints in the following symptom measure:
  • Negative symptoms will be additionally assessed using the Brief Negative Symptom Scale (BNSS).
Clinical response 4 | at inclusion; at 1-week; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to after tDCS, 1-month and 3-months endpoints in the following symptom measure:
  • Depressive symptoms will be assessed using the Calgary Depression Scale for Schizophrenia (CDSS) total score.
Clinical response 5 | at inclusion; at 1-week; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to after tDCS, 1-month and 3-months endpoints in the following symptom measure:
  • Global symptom severity and treatment response will be assessed using the Clinical Global Impressions Scale (CGI) total score.
Clinical response 6 | at inclusion; at 1-week; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to after tDCS, 1-month and 3-months endpoints in the following symptom measure:
  • Subjective experience of negative symptoms will be assessed using the Self-evaluation of Negative Symptoms (SNS) total score
Clinical response 7 | at inclusion; at 1-week; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to after tDCS, 1-month and 3-months endpoints in the following symptom measure:
  • Subjective experiences of cognitive impairment will be assessed using the self-rated Subjective Scale To Investigate Cognition in Schizophrenia (SSTICS) total score.
Outcome response 1 | at inclusion; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to 1-month and 3-months endpoints in the following general outcome measures:
  • Functional outcome will be assessed using the FROGS (Functional Remission Observatory Group in Schizophrenia) total score
Outcome response 2 | at inclusion; at 1-month follow-up; at 3-months follow-up
  Changes from baseline to 1-month and 3-months endpoints in the following general outcome measures:
  • Quality of life will be assessed by the Schizophrenia Quality of Life Questionnaire Short Form (S-QoL 18) total score
Tolerance 1 | at 1-week
  Score after the last tDCS session in the following tolerance measure:
  • tDCS-AEQ (Adverse Effects Questionnaire)
Tolerance 2 | at 1-week
  Score after the last tDCS session in the following tolerance measure:
  • VAMS (Visual Analogue Mood Scale)
Response marker 1 | at inclusion
  The differences at baseline in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • correlations (z-scores) between left prefrontal and temporal cortical areas (i.e., areas stimulated with tDCS) measured with resting-state functional Magnetic Resonance Imaging (MRI).
Response marker 2 | at inclusion
  The differences at baseline in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • spectral power (dB) in gamma frequency (40-Hz) during specific auditory paradigms (auditory steady-state, oddball, tone-matching) measured with electroencephalography (EEG).
Response marker 3 | at inclusion
  The differences at baseline in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • inter-assay coherence (%) in gamma frequency (40-Hz) during specific auditory paradigms (auditory steady-state, oddball, tone-matching) measured with electroencephalography (EEG).
Response marker 4 | at inclusion
  The differences at baseline in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • GABA and Glutamate levels (mM) within left prefrontal and temporal cortical areas measured with resting-state Magnetic Resonance Spectroscopy (MRS)
Response marker 5 | at inclusion
  The differences at baseline in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • radiotracer binding potential on GABA-A receptors (Binding Potential) within left prefrontal and temporal cortical areas measured with resting-state [11C]flumazenil Positron Emission Tomography MRI (PET-MRI).
Response predictor 1 | at inclusion; at 1-month follow-up
  Changes from baseline to 1-month in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • correlations (z-scores) between left prefrontal and temporal cortical areas (i.e., areas stimulated with tDCS) measured with resting-state functional Magnetic Resonance Imaging (MRI).
Response predictor 2 | at inclusion; at 1-month follow-up
  Changes from baseline to 1-month in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • spectral power (dB) in gamma frequency (40-Hz) during specific auditory paradigms (auditory steady-state, oddball, tone-matching) measured with electroencephalography (EEG).
Response predictor 3 | at inclusion; at 1-month follow-up
  Changes from baseline to 1-month in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • inter-assay coherence (%) in gamma frequency (40-Hz) during specific auditory paradigms (auditory steady-state, oddball, tone-matching) measured with electroencephalography (EEG).
Response predictor 4 | at inclusion; at 1-month follow-up
  Changes from baseline to 1-month in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • GABA and Glutamate levels (mM) within left prefrontal and temporal cortical areas measured with resting-state Magnetic Resonance Spectroscopy (MRS)
Response predictor 5 | at inclusion; at 1-month follow-up
  Changes from baseline to 1-month in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • GABA and Glutamate levels (mM) within left prefrontal and temporal cortical areas measured with resting-state Magnetic Resonance Spectroscopy (MRS)
Response predictor 6 | at inclusion; at 1-month follow-up
  Changes from baseline 1-month in the following early auditory processing (EAP) measure between patients with cognitive improvement and patients without cognitive improvement after active tDCS:
  • radiotracer binding potential on GABA-A receptors (Binding Potential) within left prefrontal and temporal cortical areas measured with resting-state [11C]flumazenil Positron Emission Tomography MRI (PET-MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Clément DONDÉ, Principal Investigator — CHU Grenoble Alpes
Locations (4):
- France (4):
  - CHU Grenoble Alpes, La Tronche, Auvergne-Rhône-Alpes
  - CH Alpes-Isère, Saint-Égrève, Auvergne-Rhône-Alpes
  - CH Le Vinatier, Bron
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Yes
The data will be available from the principal investigator to other study investigators or scientists upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Paper CRFs will be kept in locked files at the study sites for 15 years. In all study-related documents, participants will appear only in the form of an ID code to ensure confidentiality. All members of the research staff who will have direct access to the data before, during and after the trial will be bound to strict confidentiality rules and will not be allowed to disclose and personal or medical information.
Access Criteria: The data will be available from the principal investigator to other study investigators or scientists upon reasonable request.

REFERENCES:
- [Derived] Donde C, Bastin J, Pouchon A, Costes N, Fakra E, Galvao F, Gay A, Haesebaert F, Lamalle L, Merida I, Rigon M, Schneider F, Tropres I, Brunelin J, Polosan M. Efficacy and auditory biomarker analysis of fronto-temporal transcranial direct current stimulation (tDCS) in targeting cognitive impairment associated with recent-onset schizophrenia: study protocol for a multicenter randomized double-blind sham-controlled trial. Trials. 2023 Feb 24;24(1):141. doi: 10.1186/s13063-023-07160-z. PMID 36829240